CLINICAL TRIAL: NCT04611360
Title: Effects of Anodal Transcranial Direct Current Stimulation on Mobility and Balance in Post Stroke Patients.
Brief Title: Anodal Transcranial Direct Current Stimulation on Mobility and Balance in Post Stroke Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rec/00502 Sundus Akhtar
Record Dates: First submitted 2020-10-26; First posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Stroke
Keywords: Balance; Stroke; Anodal Transcranial Direct Current Stimulation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anodal Transcranial Direct Current Stimulation Group (Experimental): Anodal Transcranial Direct Current Stimulation and Conventional training exercises
  Interventions: Other: Anodal Transcranial Direct Current Stimulation Group
- Conventional Training Exercises Group (Active Comparator): Conventional Training Exercises : Bridging,Sitting: weight-bearing, Standing: weight-bearing, Sit to stand, Squat exercises and Tandem walk
  Interventions: Other: Conventional Training Exercises Group

INTERVENTIONS:
Other: Anodal Transcranial Direct Current Stimulation Group — Experimental group were received anodal transcranial direct current stimulation and conventional training exercises for 3 days a weeks for 6 consecutive weeks on alternate days.
  Anodal tDCS were given through:
  i. Anodal electrode:It has been placed over primary motor cortex(ipsilesional) ii. Cathodal electrode: It has been above contralateral eye. iii. Intensity: 2mA iv Density: 0.07C/cm2 iv. Duration:20 min vi Rectangular electrodes(25cm2 ) inserted in saline soaked sponge used
  Arms: Anodal Transcranial Direct Current Stimulation Group
Other: Conventional Training Exercises Group — Conventional physical exercises were given for 3 days a week on alternate days upto 6 weeks. It includes: progressive Conventional Training Exercises : From Bridging,Sitting: weight-bearing, Standing: weight-bearing, Sit to stand, Squat exercises and Tandem walk.
  Arms: Conventional Training Exercises Group

SUMMARY:
To determine the effects of anodal transcranial direct current stimulation on mobility and balance in post stroke patients.

DETAILED DESCRIPTION:
Stroke is characterised as sudden onset of neurological dysfunction of central anxious framework that contain cerebral infarction, intra cranial haemorrhage & subarachnoid haemorrhage. Around the globe stroke is the chief cause of incapacity and passing.

The trans-cranial direct current stimulations (tDCS) could be a non-invasive,low cost and capable brain stimulator utilised within the treatment of brain disorders.Two modes of tDCS is utilised is stroke patients,anodal stimulation (increased in excitability) of the lesional half of the globe and cathodal stimulation (decreased in excitability) of the contralesional hemisphere. The transcranial direct current stimulation induced polarity-dependent changes in membrane excitability, with Anodal-tDCS causing depolarisation and cathodal-tDCS causing hyper polarization of membrane potential in neurons of the stimulated area.

The role of Trans-cranial Direct Current Stimulation as a catalyst of recovery in stroke population and found that it's a safe,portable,non invasive brain stimulation technique. T-DCS is able to modulate the excitability of specified brain areas by varying the neuronal membrane potentials that based on the polarity of the current transmitted through the scalp via sponge electrodes. Trans-cranial direct current stimulation is clinically potential for use in stroke recovery because of its ease of use, non invasive-ness and safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with both ischemic and hemorrhagic stroke
* Subacute and chronic stroke patients(onset of stroke from 3 months to 1 year)
* Ambulatory stroke survivors were included who met the criteria of Modified Rankin Scale between 1 and 3

Exclusion Criteria:

* Patients with Modified Rankin Scale of 0 and 4-6.
* Brain tumors
* Cognitive impaired
* Known case of seizures
* Metal implant, head injury etc and other disorders which contraindicate the application of anodal transcranial direct current stimulations.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale | 6 week
  It is commonly used for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other neurological disorders.The scale runs from 0-6,running from perfect no symptoms to death.The inter rater reliability of Modified Rankin Scale (MRS) for stroke is (0.95)
Dynamic Gait Index | 6 week
  Dynamic Gait Index (DGI) was to evaluate functional stability in older people and to evaluate their risk of falling.Its a 4 point ordinal scale,ranging from 0-3, "0" indicates the lowest level of function and "3" indicates the highest level of function.The inter rater reliability of DGI for stroke is (0.96)
10 Meter Walk Test | 6 week
  It is to be used for gait speed assesment.According this,individual walk without assistance 10 meters and the time is measured for the intermediate 6 meters. The reliability of 10 meter walk test is (0.97)
Fugl Meyer function test: | 6 week
  Fugl Meyer Function (FMA) is used to assess voluntary movements,reflex activity,grasping and co-ordination of affected limb in stroke.It contain 33 task with a scale of 0-2 with maximum scoring of 66.The reliability of FMA scale is (0.95-1)

CONTACTS AND LOCATIONS:
Overall Officials: Mirza Obaid Baig, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rossi C, Sallustio F, Di Legge S, Stanzione P, Koch G. Transcranial direct current stimulation of the affected hemisphere does not accelerate recovery of acute stroke patients. Eur J Neurol. 2013 Jan;20(1):202-4. doi: 10.1111/j.1468-1331.2012.03703.x. Epub 2012 Mar 26. PMID 22448901
- [Background] Iosa M, Morone G, Fusco A, Bragoni M, Coiro P, Multari M, Venturiero V, De Angelis D, Pratesi L, Paolucci S. Seven capital devices for the future of stroke rehabilitation. Stroke Res Treat. 2012;2012:187965. doi: 10.1155/2012/187965. Epub 2012 Dec 13. PMID 23304640
- [Background] Fusco A, Iosa M, Venturiero V, De Angelis D, Morone G, Maglione L, Bragoni M, Coiro P, Pratesi L, Paolucci S. After vs. priming effects of anodal transcranial direct current stimulation on upper extremity motor recovery in patients with subacute stroke. Restor Neurol Neurosci. 2014;32(2):301-12. doi: 10.3233/RNN-130349. PMID 24398722